CLINICAL TRIAL: NCT06962280
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Long-Term Safety of Tirzepatide Once Weekly Compared to Placebo in Adults With Type 1 Diabetes and Obesity or Overweight
Brief Title: A Long-Term Study of Tirzepatide (LY3298176) in Adults With Type 1 Diabetes and Obesity or Overweight
Acronym: SURPASS-T1D-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27340; 2024-519685-51-00 (EU CTIS Number); I8F-MC-GPJD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-06; First posted 2025-05-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive tirzepatide subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to find out how well and how safely tirzepatide works long-term in adults who have type 1 diabetes and obesity or overweight. Participation in the study will last about 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 diabetes and on insulin treatment for at least one year prior to screening
* Have an HbA1c value of 7.0% to 10.5% inclusive, at screening
* Have a body mass index (BMI) of ≥25 kilograms per square meter (kg/m2) at screening
* Are of stable weight for at least 90 days prior to screening and agree to not start an intensive diet or exercise program during the study

Exclusion Criteria:

* Have experienced two or more events requiring hospitalization due to poor glucose control (hyperglycemia or (diabetic ketoacidosis (DKA)) during the period of 180 days prior to screening and until randomization.
* Have experienced one or more events of severe hypoglycemia during the period of 90 days prior to screening and until randomization.
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have had chronic or acute pancreatitis
* Have used any weight loss drugs or alternative remedies, including herbal or nutritional supplements, within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Change from Baseline in HbA1c | Baseline, Week 72
Percentage of Time Continuous Glucose Monitor (CGM) Glucose Values are Between 70 and 180 milligrams per deciliter (mg/dL) (3.9 and 10.0 millimoles per liter (mmol/L)) Inclusive, Per Day | Within 30 days prior to Week 40, Within 30 days prior to Week 72
Change from Baseline in Body Weight | Baseline, Week 40, Week 72
Percent Change from Baseline in Body Weight | Baseline, Week 40, Week 72
Percentage of Participants with ≥5% Body Weight Reduction | Baseline, Week 40, Week 72
Percentage of Participants with ≥10% Body Weight Reduction | Baseline, Week 40, Week 72
Percentage of Participants with ≥15% Body Weight Reduction | Baseline, Week 40, Week 72
Change from Baseline in Waist Circumference | Baseline, Week 40, Week 72
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 40, Week 72
Percent Change from Baseline in Fasting Triglycerides | Baseline, Week 40, Week 72
Percent Change from Baseline in Fasting Non-High-Density Lipoprotein (non-HDL) Cholesterol | Baseline, Week 40, Week 72
Percent Change from Baseline in Total Daily Insulin Dose | Baseline, Week 40, Week 72
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 40, Week 72
Change from Baseline in EQ-5D-5L | Baseline, Week 40, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (79):
- United States (18):
  - Kaiser Permanente Bonita Medical Offices, Bonita, California
  - AMCR Institute, Escondido, California
  - Mary & Dick Allen Diabetes Center, Newport Beach, California
  - University Clinical Investigators, Inc., Tustin, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Las Vegas Endocrinology, Henderson, Nevada
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
- Argentina (8):
  - Buenos Aires Macula S.A, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Centro Diabetológico Dr. Waitman, Córdoba
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Instituto Médico Catamarca IMEC, Rosario
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
- Brazil (8):
  - Centro de Pesquisa Clinica do Brasil, Brasília
  - Centro de Pesquisa Sao Lucas, Campinas
  - Quanta Diagnóstico e Terapia, Curitiba
  - Cendi - Endocrinologia e Diabetes, Goiânia
  - Instituto da Crianca com Diabetes, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Canada (5):
  - Endocrinologie Oasis, Montreal
  - Centricity Research Ottawa LMC Endocrinology, Ottawa
  - Centre de Recherche Saint-Louis, Sherbrooke
  - TLC Diabetes and Endocrinology, Surrey
  - Care Access - Cape Breton, Sydney
- Czechia (6):
  - INTENDIA klinika s.r.o., Chrudim III
  - AIDIN VK s.r.o., Hranice
  - MUDr. Tomas Edelsberger, Krnov
  - Diabetologicke centrum s.r.o., Olomouc
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - ResTrial s.r.o., Prague
- France (8):
  - Centre Hospitalier Universitaire - Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hôtel-Dieu du Creusot - site Harfleur, Le Creusot
  - Hôpital de la Conception, Marseille
  - Assistance Publique Hôpitaux de Paris - Groupe Hospitalier 10e - Hôpital Lariboisière, Paris
  - CHU Rangueil, Toulouse
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux
- Greece (4):
  - Athens Medical Center, Athens
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Mexico (9):
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - CEINV Salud, Monterrey
  - Clínica García Flores SC, Monterrey
  - Consultorio Médico de Endocrinología y Pediatría, Puebla City
  - Medsal Centro Médico, Tampico
- Romania (8):
  - CMI DNBM Dr. Pop Lavinia, Baia Mare
  - Mariodiab Clinic, Brasov
  - Centrul medical DiabNutriMed, Bucharest
  - Diabet Med, Bucharest
  - Sanamed Hospital, Bucharest
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Rinart Diab SRL, Târgovişte
- Spain (5):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Long-Term Study of Tirzepatide (LY3298176) in Adults With Type 1 Diabetes and Obesity or Overweight (SURPASS-T1D-2) — https://trials.lilly.com/en-US/trial/605555